CLINICAL TRIAL: NCT04878536
Title: Efficacy Testing of Collagen Drink
Brief Title: Efficacy Testing of Collagen Elixir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-042-B
Record Dates: First submitted 2021-05-06; First posted 2021-05-07 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Blank
- Collagen drink (Experimental)
  Interventions: Dietary Supplement: Collagen drink

INTERVENTIONS:
Dietary Supplement: Collagen drink — Testing product
  Other Names: Isagenix-Collagen Elixir
  Arms: Collagen drink
Dietary Supplement: Blank — Placebo drink
  Arms: Placebo drink

SUMMARY:
To assess Isagenix-Collagen Elixir on skin condition improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 20 years old

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* Patients with diseases of the skin, liver, kidney.
* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Received facial laser therapy, chemical peeling or UV overexposure in the past 4 weeks.
* Constant drug use
* Participated cosmetic product human study in the past 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
The change of skin wrinkles | Change from Baseline skin wrinkles at 4 weeks
  VISIA Complexion Analysis System was utilized to measure skin wrinkles. Units: arbitrary units
The change of skin texture | Change from Baseline skin texture at 4 weeks
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin collagen density | Change from Baseline skin collagen density at 4 weeks
  DermaLab® Series SkinLab Combo was utilized to measure skin pores. Units: arbitrary units
The change of skin elasticity | Change from Baseline skin elasticity at 4 weeks
  Soft Plus was utilized to measure skin elasticity. Units: arbitrary units
The change of MMP-1 of blood | Change from Baseline MMP-1 at 4 weeks
  Venous blood was sampled to measure MMP-1
The change of TIMP-1 of blood | Change from Baseline TIMP-1 at 4 weeks
  Venous blood was sampled to measure TIMP-1

SECONDARY OUTCOMES:
The change of skin melanin index | Change from Baseline skin melanin index at 4 weeks
  Soft Plus was utilized to measure skin melanin index. Units: arbitrary units
The change of skin L* value | Change from Baseline L* value at 4 weeks
  Chroma Meter MM500 was utilized to measure skin L* value. Units: arbitrary units, 0-100
The change of skin moisture | Change from Baseline skin moisture at 4 weeks
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
The change of skin spots | Change from Baseline skin spots at 4 weeks
  VISIA Complexion Analysis System was utilized to measure skin spots. Units: arbitrary units
The change of skin UV spots | Change from Baseline skin UV spots at 4 weeks
  VISIA Complexion Analysis System was utilized to measure skin UV spots. Units: arbitrary units
The change of skin brown spots | Change from Baseline skin brown spots at 4 weeks
  VISIA Complexion Analysis System was utilized to measure skin brown spots. Units: arbitrary units
The change of TNF-α of blood | Change from Baseline TNF-α at 4 weeks
  Venous blood was sampled to measure TNF-α
The change of IL-10 of blood | Change from Baseline IL-10 at 4 weeks
  Venous blood was sampled to measure IL-10
The change of SOD-RBC of blood | Change from Baseline SOD-RBC at 4 weeks
  Venous blood was sampled to measure SOD-RBC
The change of f-thiols of blood | Change from Baseline f-thiols at 4 weeks
  Venous blood was sampled to measure f-thiols
The change of t-GSH of blood | Change from Baseline t-GSH at 4 weeks
  Venous blood was sampled to measure t-GSH
The change of GST-RBC of blood | Change from Baseline GST-RBC at 4 weeks
  Venous blood was sampled to measure GST-RBC
The change of MDA of blood | Change from Baseline MDA at 4 weeks
  Venous blood was sampled to measure MDA
The change of blood total antioxidant capacity (TAC) | Change from Baseline TAC at 4 weeks
  Venous blood was sampled to measure concentrations of TAC

OTHER OUTCOMES:
The change of total cholesterol of blood | Change from Baseline total cholesterol at 4 weeks
  Venous blood was sampled to measure total cholesterol
The change of triglyceride of blood | Change from Baseline triglyceride at 4 weeks
  Venous blood was sampled to measure triglyceride
The change of SGOT of blood | Change from Baseline SGOT at 4 weeks
  Venous blood was sampled to measure SGOT
The change of SGPT of blood | Change from Baseline SGPT at 4 weeks
  Venous blood was sampled to measure SGPT
The change of BUN of blood | Change from Baseline BUN at 4 weeks
  Venous blood was sampled to measure BUN
The change of creatinine of blood | Change from Baseline creatinine at 4 weeks
  Venous blood was sampled to measure creatinine
The change of uric acid of blood | Change from Baseline uric acid at 4 weeks
  Venous blood was sampled to measure uric acid

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy & Science, Tainan, Taiwan